CLINICAL TRIAL: NCT02438748
Title: The Role of Biological Stress Markers in Predicting Treatment Response to Repetitive Transcranial Magnetic Stimulation in Major Depressive Disorder
Brief Title: Biological Markers of Treatment Response to Repetitive Transcranial Magnetic Stimulation for Depression
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: B2014:102
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Oxidative Stress
Keywords: Oxidized Phosphatidylcholines; Oxylipins
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10ml of blood will be extracted at each collection. Patients will give two samples. Controls will give one sample. Following collection, blood samples will be spun to separate and extract plasma. The amount of oxidized phosphatidylcholines in the plasma will then be quantified.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Individuals undergoing Repetitive Transcranial Magnetic Stimulation treatment for major depressive disorder.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Controls: Healthy age-, and sex-matched control individuals.

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — A non-invasive method of brain stimulation.
  Groups: Patients

SUMMARY:
The main objective of this study is to determine whether biological stress markers (Oxidized Phosphatidylcholines and Oxylipins) in the blood can be used to predict the efficacy of rTMS in the treatment of major depressive disorder (MDD). It is our goal to identify biomarkers that may be used to determine which patients will benefit from rTMS treatment. A second objective of this study is to measure any changes in stress markers that occur across the course of rTMS therapy.

DETAILED DESCRIPTION:
250 patients who have been prescribed repetitive transcranial magnetic stimulation (rTMS) therapy for the treatment of major depressive disorder will be recruited for this study. Prior to undergoing rTMS, patients will give a small blood sample. An additional blood sample will be given upon completion of rTMS treatment. 60 healthy control individuals will also be recruited to provide a one-time blood sample for comparison. Control individuals will not receive rTMS treatment.

Blood samples will be analysed for levels of Oxidized Phosphatidylcholines and Oxylipins. The investigators wish to determine whether there is a difference in the pre-treatment levels of stress markers between individuals who ultimately respond to rTMS and those who do not. Additionally, the investigators wish to determine whether there is a change in stress markers as a result of rTMS treatment.

ELIGIBILITY:
Patient Inclusion Criteria:

* Patients with a major depressive episode
* Not actively receiving psychotherapy

Patient Exclusion Criteria:

* History of a psychotic episode
* History of neurological illness
* Head injury
* Active alcohol or substance abuse
* History of a seizure disorder
* Pregnant

Control Subject Exclusion Criteria:

* History of depression or psychiatric illness
* History of a psychotic episode
* History of neurological illness
* Head injury
* Active alcohol or substance abuse
* History of a seizure disorder
* Pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 250 patients with Major Depressive Disorder who have been deemed eligible for rTMS treatment. Eligible persons will be identified by a psychiatrist from among patients at the outpatient Neuromodulation and Neuropsychiatric Unit at St Boniface Hospital. 60 healthy control individuals.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2015-05; Primary Completion 2022-01 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Change in Oxidized Phosphatidylcholines in plasma | 3 weeks
  Change in Oxidized Phosphatidylcholine levels in blood plasma pre- and post-repetitive transcranial magnetic stimulation (rTMS) treatment for depression.

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Modirrousta, MD PhD FRCPC, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada